CLINICAL TRIAL: NCT00810160
Title: Phase 1A Study of Impact of Oligosaccharides and Bifidobacteria on the Intestinal Microflora of Premature Infants
Brief Title: The Impact of Oligosaccharides and Bifidobacteria on the Intestinal Microflora of Premature Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 243213; R01HD059127 (NIH); HD059127-01 (Other: UC Davis)
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Fecal Microflora in the Formula Fed Premature Infant
Keywords: probiotic; prebiotic; oligosaccharides; GOS; galacto oligosaccharides; Bifidobacterium infantis; Bifidobacterium animalis
MeSH Terms: interventions — bificin C6165, Bifidobacterium animalis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Permeate
  Interventions: Dietary Supplement: ProlactPlus
- 2 (Active Comparator): GOS
  Interventions: Dietary Supplement: GOS galacto-oligosaccharides
- 3 (Active Comparator): Bifidobacterium infantis
  Interventions: Dietary Supplement: Bifidobacterium infantis
- 4 (Active Comparator): Bifidobacterium animalis
  Interventions: Dietary Supplement: Bifidobacterium animalis

INTERVENTIONS:
Dietary Supplement: ProlactPlus — Group 1 infants will be fed a concentration of Permeate mixed with formula. The ProlactPlus will be increased each week as follows: week 1 95:5 (formula:ProlactPlus), week 2 90:10, week 3 85:15, week 4 80:20, and week 5 75:25. Caloric content is roughly as follows: week 1 21 cal/oz, week 2 22 cal/oz, week 3 23 cal/oz, week 4 24 cal/oz, and week 5 25 cal/oz.
  Other Names: human milk oligosaccharides
  Arms: 1
Dietary Supplement: GOS galacto-oligosaccharides — Group 2 infants will have their formula supplemented with galacto-oligosaccharides (GOS) for each feeding as follows: week 1 0.25 g/dL, week 2 0.5 g/dL, week 3 1.0 g/dL, week 4 1.5 g/dL, and week 5 2.0 g/dL.
  Other Names: galacto-oligosaccharides
  Arms: 2
Dietary Supplement: Bifidobacterium infantis — Group 3 infants will have their formula supplemented with B. infantis twice daily increasing the dose each week as follows: week 1 5x107, week 2 1.5x108, week 3 4.5x108, week 4 1.4x109, and week 5 4.2x109.
  Other Names: bifidobacteria; B. infantis
  Arms: 3
Dietary Supplement: Bifidobacterium animalis — Group 4 infants will have their formula supplemented with B. animalis twice daily increasing the dose each week as follows: week 1 5x107, week 2 1.5x108, week 3 4.5x108, week 4 1.4x109, and week 5 4.2x109.
  Other Names: B. animalis; bifidobacteria
  Arms: 4

SUMMARY:
The purpose of this study is to see whether dietary supplements can change the germs in the intestines of premature infants to be more like those of healthy breast fed term babies.

DETAILED DESCRIPTION:
To determine the optimum dose and optimum dietary supplement to promote a fecal microflora in the formula fed premature infant that is similar to that of the term breast fed infant (a predominance of bifidobacteria). In the initial phase of this trial, 30 premature infants will be randomly assigned to receive increasing doses of one of four dietary supplements: Permeate (a pasteurized human milk concentrate containing human milk oligosaccharides processed by Prolacta), GOS (galacto-oligosaccharides manufactured by Friesland foods), Bifidobacterium infantis or Bifidobacterium animalis. Weekly stool specimens will be examined by PCR to determine content of bifidobacteria and total bacteria. This study is limited to formula fed infants in order to avoid the confounding effects of the human milk oligosaccharides in breast milk. An additional 12 human milk fed infants will be enrolled and will have their diet supplemented with ProlactPlus (a pasteurized human milk concentrate containing humna milk oligosaccharides) or powdered human milk fortifier for comparison

ELIGIBILITY:
Inclusion Criteria:

* Born in or transferred to UCDMC within the first two weeks of life. Birth weight less than 1500 grams. Gestational age less than 33 completed weeks. Exclusively formula fed.

Exclusion Criteria:

* Gastrointestinal or cardiac anomalies.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
To determine the optimum dose and optimum dietary supplement to promote a fecal microflora in the formula fed premature infant that is similar to that of the term breast fed infant (a predominance of bifidobacteria). | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Underwood, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Derived] Underwood MA, Kalanetra KM, Bokulich NA, Lewis ZT, Mirmiran M, Tancredi DJ, Mills DA. A comparison of two probiotic strains of bifidobacteria in premature infants. J Pediatr. 2013 Dec;163(6):1585-1591.e9. doi: 10.1016/j.jpeds.2013.07.017. Epub 2013 Aug 29. PMID 23993139